CLINICAL TRIAL: NCT00316914
Title: A Phase III Randomized, Placebo-Controlled, Double-Blind Study of Intravenous Calcium/Magnesium to Prevent Oxaliplatin-Induced Sensory Neurotoxicity
Brief Title: Calcium Gluconate and Magnesium Sulfate in Preventing Neurotoxicity Caused By Oxaliplatin in Patients Receiving Combination Chemotherapy for Stage II, Stage III, or Stage IV Colorectal Cancer That Has Been Completely Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N04C7; NCCTG-N04C7; CDR0000471238 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Results first posted 2013-03-25 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer; Neurotoxicity
Keywords: neurotoxicity; stage II colon cancer; stage III colon cancer; adenocarcinoma of the colon; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; stage IV colon cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Neurotoxicity Syndromes; Colonic Neoplasms; Rectal Neoplasms | interventions — Calcium Gluconate; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ca/Mg (Experimental): Patients receive calcium gluconate (Ca) and magnesium sulfate (Mg) IV over 30 minutes immediately before and after each oxaliplatin administration (once every 2 weeks) of their assigned chemotherapy regimen.
  Interventions: Drug: calcium gluconate; Drug: magnesium sulfate
- Placebo (Placebo Comparator): Patients receive a placebo IV over 30 minutes immediately before and after each oxaliplatin administration (once every 2 weeks) of their assigned chemotherapy regimen.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: calcium gluconate — Given IV
  Arms: Ca/Mg
Drug: magnesium sulfate — Given IV
  Arms: Ca/Mg
Other: placebo — Given IV
  Arms: Placebo

SUMMARY:
RATIONALE: Calcium gluconate and magnesium sulfate may prevent or lessen neurotoxicity caused by oxaliplatin. It is not yet known whether calcium gluconate and magnesium sulfate are more effective than a placebo in preventing neurotoxicity caused by oxaliplatin in patients receiving combination chemotherapy.

PURPOSE: This randomized phase III trial is studying calcium gluconate and magnesium sulfate to see how well they work compared to a placebo in preventing neurotoxicity caused by oxaliplatin in patients receiving combination chemotherapy for stage II, stage III, or stage IV colorectal cancer that has been completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether calcium gluconate and magnesium sulfate (CaMg) infusions can prevent or ameliorate chronic, cumulative oxaliplatin-induced neurotoxicity in patients receiving FOLFOX combination chemotherapy for stage II, III or IV colorectal cancer.
* Determine whether CaMg infusions can increase the cumulative oxaliplatin doses that can be delivered without chronic neurotoxicity.
* Determine whether CaMg infusions can ameliorate the acute neuropathy associated with oxaliplatin.
* Determine whether CaMg infusions cause any adverse events.
* Investigate whether CaMg infusions influence quality of life, fatigue, and activities of daily living of these patients.
* Determine if polymorphisms in the GSTP1 gene predict early onset of oxaliplatin-induced neurotoxicity.

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are stratified according to age (< 65 vs > 65), gender, and chemotherapy regimen (FOLFOX4 vs modified FOLFOX6). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and after each oxaliplatin administration (once every 2 weeks) of their assigned chemotherapy regimen.
* Arm II: Patients receive a placebo IV over 30 minutes immediately before and after each oxaliplatin administration (once every 2 weeks) of their assigned chemotherapy regimen.

In both arms, treatment continues until chemotherapy is discontinued (approximately 6 months).

Patients complete quality of life questionnaires on day 1, a symptom experience diary on days 2-5 of their chemotherapy regimen, and questionnaires at 1 and 3 months after completion of study treatment.

Blood samples are collected at baseline and tested for the GSTP1 gene.

After completion of study treatment, patients are followed for at least 3 months.

PROJECTED ACCRUAL: A total of 300 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Stage II disease
  * Stage III disease
  * Stage IV disease (completely resected with no evidence of residual tumor)
* Must have undergone curative resection for stage II or III disease
* Scheduled to receive 6 months of adjuvant treatment with either of the following FOLFOX chemotherapy regimens:

  * FOLFOX4, comprising leucovorin calcium, fluorouracil, and oxaliplatin (2-week course)
  * Modified FOLFOX6, comprising high-dose leucovorin calcium, high-dose fluorouracil, and oxaliplatin (2-week course)

PATIENT CHARACTERISTICS:

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* WBC ≥ 3,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Calcium normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No pre-existing peripheral neuropathy of any grade
* No hypercalcemia
* No concurrent heart block or a history of heart block
* No other medical condition that, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
* No family history of a genetic/familial neuropathy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior treatment with neurotoxic chemotherapy such as oxaliplatin, cisplatin, taxanes, or vinca alkaloids
* Concurrent use of bevacizumab or cetuximab in combination with FOLFOX as part of a clinical trial or clinical practice are allowed
* No concurrent digitalis medication
* No concurrent digoxin
* No concurrent treatment with anticonvulsants such as carbamazepine, phenytoin, or valproic acid
* No other concurrent neurotropic agents such as gabapentin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Grothey, MD, Study Chair — Mayo Clinic
Locations (14):
- United States (14):
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota

REFERENCES:
- [Result] Grothey A, Nikcevich DA, Sloan JA, Kugler JW, Silberstein PT, Dentchev T, Wender DB, Novotny PJ, Chitaley U, Alberts SR, Loprinzi CL. Intravenous calcium and magnesium for oxaliplatin-induced sensory neurotoxicity in adjuvant colon cancer: NCCTG N04C7. J Clin Oncol. 2011 Feb 1;29(4):421-7. doi: 10.1200/JCO.2010.31.5911. Epub 2010 Dec 28. PMID 21189381
- [Result] Nikcevich DA, Grothey A, Sloan JA, et al.: Effect of intravenous calcium and magnesium (IV CaMg) on oxaliplatin-induced sensory neurotoxicity (sNT) in adjuvant colon cancer: results of the phase III placebo-controlled, double-blind NCCTG trial N04C7. [Abstract] J Clin Oncol 26 (Suppl 15): A-4009, 2008.
- [Derived] Pachman DR, Qin R, Seisler DK, Smith EM, Beutler AS, Ta LE, Lafky JM, Wagner-Johnston ND, Ruddy KJ, Dakhil S, Staff NP, Grothey A, Loprinzi CL. Clinical Course of Oxaliplatin-Induced Neuropathy: Results From the Randomized Phase III Trial N08CB (Alliance). J Clin Oncol. 2015 Oct 20;33(30):3416-22. doi: 10.1200/JCO.2014.58.8533. Epub 2015 Aug 17. PMID 26282635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One-hundred and four (104) participants were recruited between January 2006 and June 2007 from 20 North Central Cancer Treatment Group (NCCTG) member sites.
Pre-assignment Details: Two participants in Calcium/Magnesium arm canceled prior to study medication begins. These two participants were excluded from all analysis.
Period: Overall Study
Arm/Group | Ca/Mg | Placebo
Started | 50 | 52
Completed | 17 | 16
Not Completed | 33 | 36
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Adverse Event | 8 | 7
Not completed — Other Problems | 6 | 11
Not completed — Missing end of treatment documentation | 14 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ca/Mg | Placebo | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Customized [Number; unit: Participants]
  <65 | 33 | 33 | 66
  >=65 | 17 | 19 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 27 | 27 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 48 | 50 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 52 | 102
Regimen [Number; unit: Participants]
  FOLFOX4 (Oxaliplatin, Leucovorin, and Fluorouracil | 3 | 3 | 6
  Modified FOLFOX6 | 47 | 49 | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Oxaliplatin-induced Grade 2+ Chronic Neuropathic Adverse Event
Description: Neuropathic adverse events were assessed by Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Neurotoxicity evaluation grade: loss of deep tendon reflexes or paresthesia, including tingling, but not interfering with function (Grade 1); objective sensory alteration or paresthesia, including tingling, interfering with function, but not with activities of daily living (Grade 2); sensory alteration or paresthesia interfering with activities of daily living (Grade 3); permanent sensory losses that are disabling (Grade 4)
Time Frame: 127 days
Population: Efficacy analyses use all patients that reported at least one value after baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 50 | 52
Percentage of participants | 22 | 41
Statistical Analysis 1: Comparison: Ca/Mg vs Placebo; Comparison in Percentage of Patients With Oxaliplatin-induced Grade 2+ Chronic Neuropathic Adverse Event between Arms; Test type: Superiority or Other; p = 0.038, Chi-squared — A priori threshold for the p-value is 0.05 and there was no adjustment for multiple comparisons

2. Secondary Outcome: Time to Onset of Grade 2+ Chronic Neurotoxicity
Description: Neurotoxicity were assessed by Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
Time Frame: 127 days
Population: Includes all patients that reported at least one value after baseline.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 50 | 52
Days | NA [NA to NA] — The median and 95% confidence interval was not calculable because insufficient number of participants reached the event at the final time point for assessment. | 18.1 [15 to NA] — The upper limit of the 95% confidence interval was infinity.
Statistical Analysis 1: Comparison: Ca/Mg vs Placebo; Comparison of time to Onset of Grade 2+ Chronic Neurotoxicity between Arms; Test type: Superiority or Other; p = 0.0503, Log Rank

3. Secondary Outcome: Time to Onset of Grade 3+ Chronic Neurotoxicity
Description: Neurotoxicity was assessed by CTCAE v3.0.
Time Frame: 127 days
Population: Includes all patients that reported at least one value after baseline.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 50 | 52
Days | NA [NA to NA] — The median and 95% confidence interval was not calculable because insufficient number of participants reached the event at the final time point for assessment. | NA [NA to NA] — The median and 95% confidence interval was not calculable because insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Ca/Mg vs Placebo; Comparison of Time to Onset of Grade 3+ Chronic Neurotoxicity between Arms; Test type: Superiority or Other; p = 0.4048, Log Rank

4. Secondary Outcome: Average Duration of Chronic Neuropathic Toxicity
Description: Neuropathic adverse events were assessed by CTCAE v3.0.
Time Frame: 127 days
Population: Includes all patients that reported at least one value after baseline.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 50 | 52
days | 81 [52 to 92] | 72 [43 to 85]
Statistical Analysis 1: Comparison: Ca/Mg vs Placebo; Comparison of Average Duration of Chronic Neuropathic Toxicity between Arms; Test type: Superiority or Other; p = 0.6556, Log Rank

5. Secondary Outcome: Percentage of Patients Discontinuing Therapy for Chronic Neurotoxicity
Description: Neurotoxicity were assessed by CTCAE v3.0.
Time Frame: 127 days
Population: Includes all patients that reported at least one value after baseline.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 50 | 52
Percentage of Participants | 46 | 55.8
Statistical Analysis 1: Comparison: Ca/Mg vs Placebo; Comparison of Percentage of patients discontinuing therapy for chronic neurotoxicity between Arms; Test type: Superiority or Other; p = 0.3238, Chi-squared

6. Secondary Outcome: Average Cumulative Oxaliplatin Dose
Time Frame: 127 days
Population: Because of the early closure of this trial, no reliable data were available for this outcome.
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Average Duration of Oxaliplatin-containing Treatment
Time Frame: 127 days
Population: Because of the early closure of this trial, no reliable data were available for this outcome.
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Patients With Acute Neuropathic Adverse Event
Description: Acute neuropathic toxicities were measured using the Symptom Experience Diary and supplemental quality of life questions in the scale of 0 (no symptom) to 10 (worst symptom). The item score was reversed and transformed into 0 (low QOL) to 100 (best QOL) scale for analysis. Any score greater than 0 was considered having acute neuropathy.
Time Frame: 127 days
Population: Includes all patients that reported at least one value after baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 50 | 52
Percentage of participants | 88 | 90
Statistical Analysis 1: Comparison: Ca/Mg vs Placebo; Comparison of Percentage of Patients With Acute Neuropathic Adverse Event between Arms; Test type: Superiority or Other; p = 0.7498, Chi-squared

9. Secondary Outcome: Incidence of Calcium Magnesium (CaMg)-Induced Adverse Event
Description: Adverse Events were measured using CTCAE V3.0.
Time Frame: 127 days
Population: Analyses of adverse events includes all patients. Adverse event data is not available on one patient in Placebo arm, which leads to the total of 51 in Placebo arm for analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 50 | 51
Percentage of Participants
  Abdominal Infection | 2 | 0
  Acne NOS | 2 | 2
  Anemia | 4 | 4
  Anorexia | 4 | 2
  Clostridial Infection | 0 | 2
  Constipation | 42 | 47
  Dehydration | 2 | 6
  Diarrhea-No Colostom | 68 | 73
  Dry Skin | 0 | 2
  Erythema Multiforme | 4 | 0
  Fatigue | 10 | 25
  Hypercalcemia | 0 | 2
  Hyperglycemia | 2 | 0
  Hypermagnesemia | 14 | 18
  Hypersensitivity | 6 | 0
  Hypokalemia | 4 | 2
  Hypomagnesemia | 0 | 2
  Hyponatremia | 4 | 0
  Infection | 0 | 2
  Ischemia-Cerebral | 0 | 2
  Ischemia/Infarction | 2 | 0
  Laryngeal Discomfort | 0 | 2
  Leukopenia | 6 | 10
  Muscle Weakness | 2 | 0
  Myalgia | 4 | 0
  Nausea | 60 | 71
  Neuro-motor | 4 | 4
  Neuro-sensory | 2 | 12
  Neutropenia | 18 | 33
  Oral cavity MS CE | 2 | 0
  Pain-Abdominal | 0 | 8
  Pain-Chest | 0 | 2
  Pain-Headache | 0 | 4
  Rash/Desquamation | 4 | 0
  Skin Rxn-Hand/Foot | 4 | 2
  Stomatitis | 2 | 2
  Taste | 2 | 2
  Thrombocytopenia | 2 | 2
  Thrombosis | 6 | 4
  Urticaria | 0 | 2
  Vasc Access Complication | 2 | 0
  Vomiting | 34 | 33

10. Secondary Outcome: Percentage of Patients Experiencing Impact on Activities of Daily Living (ADL)
Description: Activities of daily living were measured using the Symptom Experience Diary and supplemental quality of life questions. The questionnaires' items were in the scale of 0 (no symptom) to 10 (worst symptom).
Time Frame: 127 days
Population: Data was collected but not analyzed for this outcome.
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Fatigue Score at One Month
Description: Fatigue was measured by Brief Fatigue Inventory in the scale of 0 (no fatigue) to 10 (fatigue as bad as you can imagine). The item score was reversed and transformed into 0 (low quality of life (QOL)) to 100 (best QOL) scale for analysis. Change: score at one month minus score at baseline.
Time Frame: Baseline and One month
Population: Includes all patients with at least one assessment after baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 50 | 52
units on a scale
  Fatigue NOW | 1.0 (14.96) | -2.8 (17.92)
  Fatigue USUAL | 3.1 (15.38) | -1.6 (12.81)
  Fatigue WORST | 0.0 (21.38) | -1.6 (18.41)
Statistical Analysis 1: Comparison: Ca/Mg vs Placebo; Comparison of Fatigue NOW between two arms; Test type: Superiority or Other; p = 0.2340, Kruskal-Wallis
Statistical Analysis 2: Comparison: Ca/Mg vs Placebo; Comparison of Fatigue USUAL between two arms; Test type: Superiority or Other; p = 0.2010, Kruskal-Wallis
Statistical Analysis 3: Comparison: Ca/Mg vs Placebo; Comparison of Fatigue WORST between two arms; Test type: Superiority or Other; p = 0.9364, Kruskal-Wallis

12. Secondary Outcome: Change From Baseline in Quality of Life (QOL) at One Month
Description: Quality of Life (QOL) were measured using the Symptom Experience Diary and supplemental quality of life questions. Item score range: 0 (no symptom) to 10 (worst symptom). The score was reversed and transformed into 0 (low QOL) to 100 (best QOL) scale for analysis. Change: score at one month minus score at baseline.
Time Frame: Baseline and One month
Population: Includes all patients with at least one assessment after baseline.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ca/Mg | Placebo
Number analyzed (Participants) | 50 | 52
Units on a scale
  Fatigue WORST | 0.0 (21.38) | -1.6 (18.41)
  Walking | -2.5 (11.54) | 0.2 (12.78)
  Buttoning Shirt or Tying Laces | -2.0 (9.27) | 0.4 (21.07)
  Diarrhea | -7.1 (18.43) | -10.4 (21.77)
  Constipation | -2.9 (14.87) | 0.4 (26.94)
  Abdominal Cramping | -2.5 (11.75) | 1.3 (23.46)
  Bowel Problems with Normal Activity | -3.2 (18.06) | -9.1 (19.05)
  Shortness of Breath (Week 2 - Baseline) | -0.7 (7.16) | 2.1 (22.26)
  Swallowing (Week 2 - Baseline) | -7.5 (17.56) | 2.1 (21.87)
  Numbness in Fingers, Toes (Week 2 - Baseline) | -8.3 (16.49) | -9.6 (15.74)
  Tingling in Fingers, Toes (Week 2 - Baseline) | -14.8 (21.65) | -20.4 (20.53)
Statistical Analysis 1: Comparison: Ca/Mg vs Placebo; Fatigue WORST; Test type: Superiority or Other; p = 0.9364, Kruskal-Wallis
Statistical Analysis 2: Comparison: Ca/Mg vs Placebo; Walking; Test type: Superiority or Other; p = 0.6275, Kruskal-Wallis
Statistical Analysis 3: Comparison: Ca/Mg vs Placebo; Buttoning Shirt or Tying Laces; Test type: Superiority or Other; p = 0.6988, Kruskal-Wallis
Statistical Analysis 4: Comparison: Ca/Mg vs Placebo; Diarrhea; Test type: Superiority or Other; p = 0.5124, Kruskal-Wallis
Statistical Analysis 5: Comparison: Ca/Mg vs Placebo; Constipation; Test type: Superiority or Other; p = 0.3103, Kruskal-Wallis
Statistical Analysis 6: Comparison: Ca/Mg vs Placebo; Abdominal Cramping; Test type: Superiority or Other; p = 0.8601, Kruskal-Wallis
Statistical Analysis 7: Comparison: Ca/Mg vs Placebo; Bowel Problems with Normal Activity; Test type: Superiority or Other; p = 0.2439, Kruskal-Wallis
Statistical Analysis 8: Comparison: Ca/Mg vs Placebo; Shortness of Breath (Week 2 - Baseline); Test type: Superiority or Other; p = 0.9283, Kruskal-Wallis
Statistical Analysis 9: Comparison: Ca/Mg vs Placebo; Swallowing (Week 2 - Baseline); Test type: Superiority or Other; p = 0.4715, Kruskal-Wallis
Statistical Analysis 10: Comparison: Ca/Mg vs Placebo; Numbness in Fingers, Toes (Week 2 - Baseline); Test type: Superiority or Other; p = 0.5105, Kruskal-Wallis
Statistical Analysis 11: Comparison: Ca/Mg vs Placebo; Tingling in Fingers, Toes (Week 2 - Baseline); Test type: Superiority or Other; p = 0.2181, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse events data reported as of June 2, 2008, when data is frozen for study analysis.
Description: Analyses of adverse events includes all patients.
Arm/Group | Ca/Mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/50 | 1/52
Other Adverse Events (participants affected / at risk) | 48/50 | 46/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ca/Mg (N=50) | Placebo (N=52)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ca/Mg (N=50) | Placebo (N=52)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 2 (4)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 25 (87) | 26 (75)
Diarrhea (Gastrointestinal disorders) | 37 (144) | 40 (170)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (6) | 1 (2)
Nausea (Gastrointestinal disorders) | 32 (133) | 38 (150)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 19 (39) | 19 (41)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (15) | 13 (22)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 4 (4) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 3 (8) | 6 (8)
Neutrophil count decreased (Investigations) | 9 (18) | 20 (24)
Platelet count decreased (Investigations) | 2 (2) | 3 (4)
Weight loss (Investigations) | 1 (2) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum magnesium increased (Metabolism and nutrition disorders) | 9 (21) | 10 (39)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 4 (12) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (28) | 13 (29)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (7) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 3 (7) | 3 (5)

LIMITATIONS AND CAVEATS:
Data cutoff was done after 127 days because of premature study closure and because of the protocol modification mandating that the Ca/Mg therapy be discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes